CLINICAL TRIAL: NCT06820983
Title: Evaluation of the Quality of Life of Patients With DBB With the Installation of OPEP
Acronym: EQOPEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Hôpital Armand Trousseau (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2024_843_0118
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Bronchiectasis; Quality of Life; Physiotherapy
Keywords: quality of life; Bronchiectasis; oscillating PEP devices; physiotherapy
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: adult questionnary for parents of children aged 8 to 13 — Quality of life questionnaire for parents of children aged 8 to 13
Other: Quality of life questionnaire for children aged 8 to 13 — Quality of life questionnaire for children aged 8 to 13
Other: Quality of life questionnaire for adolescents aged 14 to 17 — Quality of life questionnaire for adolescents aged 14 to 17
Other: Quality of life questionnaire for adults — Quality of life questionnaire for adults
Other: A satisfaction adherence questionnaire — A satisfaction adherence questionnaire will also be distributed to patients after several months' use of oscillating PEP

SUMMARY:
To carry out an assessment of compliance and quality of life in a population (children and adults) with DDB before and after the use of an oscillating PEP. The aim is to determine the impact of the use of oscillating PEP on the daily life of this population in particular.

ELIGIBILITY:
Inclusion Criteria:

* Children (from 8 years of age) and adults over 18 years of age with DDB who doesn't use oscillating PEP.

The study population will be clinically stable and will be seen in follow-up consultations.

Exclusion Criteria:

* Children under 8 years of age.
* Patients who use an OPEP
* Patients in the acute exacerbation phase of their DDB
* Patients who are not under regular consultation
* Patients with severe, uncontrolled co-morbidities
* Patients with cognitive or psychiatric disorders preventing proper adherence to the study protocol
* Patients taking part simultaneously in another clinical study that could interfere with the results of the OPEP study

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Variation of patient quality of life before and after OPEP installation | 18 months
  quality of life is determined by qustionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens-Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No